CLINICAL TRIAL: NCT04100343
Title: Detection of Pattern of Unusual Signs and Symptoms of Multiple Sclerosis
Brief Title: Detection of Pattern of Some Unusual Signs and Symptoms of Multiple Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmood Mohammed Yosry Abdelsatar Mohammed, Mahmood M. Yosry Abdelsatar, Assiut University
Other Study IDs: Unusual multiple sclerosis
Record Dates: First submitted 2019-09-17; First posted 2019-09-24 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Each Multiple Sclerosis patient will be submitted to Cognitive Abilities Screening Instrument (CASI), Expanded Disability Status Scale, Epowrth Sleeping Scale(ESS),Fatigue Severity Scale(FSS), Hamilton Depression Rating Scale, Hamilton Anxiety Rating Scale, Headache Disability Index, specific questionnaire based on International Headache Society (IHS) recommendations

ELIGIBILITY:
Inclusion Criteria:

1. Male or female.
2. Age:30-50 years
3. Accepting all study requirement

Exclusion Criteria:

1. comorbid patient e.g (diabetic, hypertensive.......etc )
2. opposition of the patient or their family

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will include all patients daignosed as multiple sclerosis attending at Assiut university hospital within the prescribed time
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Fatigue severity scale | 1 year
  A self-report scale of nine items about fatigue, its severity and how it affects certain activities. Answers are scored on a seven point scale where 1 = strongly disagree and 7 = strongly agree. This means the minimum score possible is nine and the highest is 63. The higher the score, the more severe the fatigue is and the more it affects the person's activities. It is simple to understand and takes an average of eight minutes to answer